CLINICAL TRIAL: NCT07168486
Title: A Phase Ia Study of Tri-specific CAR19.20.22 Chimeric Antigen Receptor (CAR) T-cells for Patients With Relapsed/Refractory B-Cell Lymphomas
Brief Title: CD19.20.22 CAR T-cells for Patients With Relapsed/Refractory B-Cell Lymphomas
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2372GCCC; HP-00107536
Record Dates: First submitted 2025-05-13; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: B-Cell Lymphoma; Diffuse Large B Cell Lymphoma (DLBCL); Primary Mediastinal Large B-cell Lymphoma (PMBCL); Follicular Lymphoma; Transformed Follicular Lymphoma (tFL); Mantle Cell Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Richter Transformation; Marginal Zone Lymphoma
Keywords: relapsed; refractory; B-Cell Malignancies; Car T-cells; Lymphodepletion
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Recurrence | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level -1 (Experimental): Autologous CAR19.20.22 T-cells, 0.75 × 10^6 cells/kg (±20%), IV infusion following fludarabine/cyclophosphamide lymphodepletion.
  Interventions: Biological: CD19.20.22 CAR T cells; Drug: Fludarabine and Cyclophosphamide
- Dose Level 0 (Experimental): Autologous CAR19.20.22 T-cells, 1.0 × 10^6 cells/kg (±20%), IV infusion following fludarabine/cyclophosphamide lymphodepletion.
  Interventions: Biological: CD19.20.22 CAR T cells; Drug: Fludarabine and Cyclophosphamide
- Dose Level 1 (Experimental): Autologous CAR19.20.22 T-cells, 2.5 × 10^6 cells/kg (±20%), IV infusion following fludarabine/cyclophosphamide lymphodepletion.
  Interventions: Biological: CD19.20.22 CAR T cells; Drug: Fludarabine and Cyclophosphamide

INTERVENTIONS:
Biological: CD19.20.22 CAR T cells — CAR19.20.22 is a type of immunotherapy known as a chimeric antigen receptor T-cells (CAR T-cells).
Drug: Fludarabine and Cyclophosphamide — Lymphodepletion with Flu-Cy prior to CAR T cell therapy

SUMMARY:
The goal of this study is to treat patients diagnosed with relapsed or refractory positive B cell lymphoma - positive for 2 or more target antigens - with CAR19.20.22 CAR T-cells.

Based on the preclinical characteristics of the LTG2950, CAR19.20.22 tri-specific CAR T-cells the Investigators have developed the following hypotheses to be tested in our phase Ia clinical trial. The Investigators hypothesize that these novel CAR T-cells will show:

* good safety and tolerability
* a high degree of efficacy
* very good persistence
* an acceptable level of exhaustion

DETAILED DESCRIPTION:
This is a phase 1a, open-label, single center study evaluating the safety and efficacy CAR19.20.22 in subjects with r/r B-cell malignancies. The study will comprise dose-escalation.

The dose-escalation will use a modified 3+3 design. Up to 12 subjects will be enrolled and treated at the sequential dose-escalation levels and evaluated. Infusion of CAR19.20.22 will be staggered to allow observations of acute and subacute toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed relapsed/refractory B cell Lymphoma. Histologies allowed: diffuse large B cell lymphoma (DLBCL), primary mediastinal large B cell lymphoma (PMBCL), Follicular Lymphoma (FL), transformed follicular lymphoma (tFL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), Richter's transformation with or without concurrent CLL, Burkitt's lymphoma.
* Relapsed or Refractory disease after two lines or more of therapy (except one or more line for MCL) including rituximab and other anti-CD20 antibodies, BTK inhibitors (Mantle Cell Lymphoma only), and anthracycline (specifically for DLBCL, PMBCL, tFL, and Burkitt's lymphoma).
* Measurable disease according to Lugano 2014 criteria for assessing FDG-PET/CT in lymphoma [2]. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy. If the only measurable disease is lymph node disease, at least 1 lymph node should be ≥ 1.5 cm.
* Two out of three target antigen expression required (IHC or flow per institutional guidelines) on the most recent biopsy available. We will analyze a tumor sample from the most recent relapse or development of refractory disease state (archival sample within <6 months) for antigen expression. Alternatively, a new biopsy will be obtained in case archival material is not available.
* Prior Auto CAR T permitted (washout 3 months)
* Prior ASCT is permitted and prior AlloSCT is permitted if off immunosuppression and no clinically significant (more than grade 1) GVHD
* Prior Allo CAR T permitted (washout 1 month, permitting hematologic parameters)
* Prior Bispecific T-Cell Engager (BiTE) permitted (washout 3 months)
* At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint (ICP) therapy and anti-CD20 mAb therapy
* At least 3 half-lives must have elapsed after any prior systemic inhibitory/stimulatory ICP or anti-CD20 mAb therapy at the time the subject is planned for leukapheresis
* ECOG 0 or 1
* Acceptable Organ and Marrow Function (supportive care is allowed per institutional standards, i.e. filgrastim, transfusion) Cardiac ejection fraction (EF) greater than or equal to 45% as determined by an echocardiogram (ECHO) or Multigated Radionuclide Angiography (MUGA) Resting O2 saturation >90% on room air Total bilirubin ≤ 1.5 mg/dL except in individuals with Gilbert's syndrome Total bilirubin ≤ 3.0 mg/dL in individuals with Gilbert's syndrome Serum alanine aminotransferase (ALT) / aspartate aminotransferase (AST) <5 times the Upper Limit of Normal (ULN) for age
* A creatinine clearance (as estimated by direct urine collection or the non-racial CKD-EPI equation) > 30 mL/min
* Subjects must have the following hematologic function parameters:

Absolute neutrophil count (ANC) > 1000/µL Absolute Lymphocyte Count > 100/µL Platelets > 50,000/µL

* Estimated life expectancy of more than 3 months independent from primary disease
* Subjects of child-bearing or child-fathering potential must be willing to use study-defined highly-effective methods birth control from the time of enrollment on this study through the study follow-up period Study-defined highly-effective methods of birth control are implants, levonorgestrel releasing intrauterine systems, medroxyprogesterone acetate depot, tubal sterilization, sexual intercourse with a vasectomised male partner only (vasectomy must be confirmed by two negative semen analyses), and ovulation inhibitory progesterone.

Exclusion Criteria:

* Unable to give informed consent
* Known history of infection with human immunodeficiency virus (HIV) or active hepatitis B (HBsAg positive), If there is a history of treated hepatitis B or hepatitis C, the viral load must be polymerase chain reaction (PCR) negative; antiviral secondary prophylaxis is required if HBsAg negative and anti-HBc positive
* Known history of infection with hepatitis C virus (anti-HCV positive) unless viral load is undetectable per quantitative PCR and/or nucleic acid testing
* Known history of active seizure or presence of seizure activities or on active anti-seizure medications within the prior 12 months
* Known history or presence of autoimmune CNS disease, such as multiple sclerosis, optic neuritis or other immunologic or inflammatory disease
* Presence of active CNS disorder that, in the judgment of the investigator, may impair the ability to evaluate neurotoxicity
* Active systemic fungal, viral or bacterial infection
* Pregnant or breast-feeding woman
* Previous or concurrent malignancy with the following exceptions:

Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 2 years prior to the study Adequately treated breast or prostate carcinoma on hormonal maintenance therapies such as Lupron or tamoxifen and in clinical remission of ≥ 2 years A primary malignancy which has been completely resected / treated with curative intent and in complete remission of ≥ 2 years History of non-neurologic autoimmune disease (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) requiring systemic immunosuppressive or systemic disease modifying agents (equivalent to > 10 mg prednisone daily) within the last 2 years

* Medical condition requiring prolonged use of systemic corticosteroids equivalent to Prednisone >10 mg/day
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 6 months of enrollment
* Concurrent radiotherapy (normal tissue sparing palliative radiotherapy allowed up to time of lymphodepletion).
* For systemic therapy, at least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed at the time of scheduled leukapheresis.
* Baseline dementia that would interfere with therapy or monitoring, determined using Immune Effector Cell-Associated Encephalopathy (ICE) Assessment at baseline.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study
* Clinical suspicion of central nervous system (CNS) lymphoma
* If the subject has history of CNS disease, then he/she must Have no signs or symptoms of active CNS disease Have no active disease on magnetic resonance imaging (MRI)- e.g. vasogenic edema; stable, post-treatment changes are acceptable.

Have no malignant cells of any type present in cerebrospinal fluid (CSF) on cytospin preparation and flow cytometry, regardless of number of white blood cells (WBCs)

* In case of cerebral vascular accident (CVA) The CVA event must be > 12 months prior to leukapheresis Any neurological deficits must be stable
* ECOG 2 or higher (unless due to lymphoma diagnosis)
* Ongoing immunosuppression for graft versus host disease treatment or prophylaxis (prior allogeneic stem cell transplant permitted)
* History of a severe hypersensitivity reaction or contraindication to any of the agents used in the study (including fludarabine and cyclophosphamide).
* Subjects of both genders who are not willing to practice highly effective birth control from the time of informed consent through 6 months after the CAR19.20.22infusion
* In the investigator's judgment, the subject is unlikely to complete all study-specific visits or procedures, including follow-up visits, or comply with the study requirements for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 [Safety and Tolerability] | From date of enrollment assessed up to 24 months
  To evaluate the safety and tolerability of CAR19.20.22 CAR T-cells
Efficacy Overall Response Rate in participants | From date of enrollment assessed up to 24 months
  Effect on the disease: Number of patients with clinical responses: Overall Survival (OS); Progression-Free Survival (PFS); Overall Response Rate (ORR)
Change in CAR19.20.22 T-cell function assessed by multicolor ELISPOT assay using CD19/CD22 protein targets. | From date of enrollment assessed up to 24 months
  Function will be assessed using in-house multicolor ELISPOT assays performed on leukapheresis product, starting T-cells, final CAR T-cell product, and post-infusion blood samples.
  To evaluate the functionality of the CAR T-cells over time using our in-house developed multicolor enzyme-linked immune absorbent spot (ELISPOT) assays using beads covered with CD19 and CD22 recombinant proteins as targets.
Persistence of CAR19.20.22 T-cells in peripheral blood measured by qPCR vector copy number and flow cytometry enumeration of CD19 and CD22 CAR-expressing T-cells." | From date of enrollment assessed up to 24 months
  PK/PD persistence will be evaluated using qPCR to quantify vector copy number and flow cytometry to enumerate CD19 and CD22 CAR-expressing T-cells.
  Pharmacokinetics/Pharmacodynamics (PK/PD) - In vivo duoCAR T-cell persistence in peripheral blood samples by qPCR to measure vector copy number or Flow Cytometry to enumerate CD19 CAR or CD22 CAR expressing T-cells.

SECONDARY OUTCOMES:
Incidence of antibodies to CAR19.20.22 T-cells | Up to 24 months
  Incidence of antibodies to CAR19.20.22 measured in serum samples (up to 24 months).
  Serum samples will be tested for anti-CAR antibody responses.
Cytokine levels in plasma post-infusion | Up to 24 months
  Cytokines such as IL-6 and IFN-γ will be measured by multiplex immunoassays.
Persistence of CAR19.20.22 T-cells | Up to 24 months
  Enumeration of CAR T-cells from blood samples using flow cytometry.
Phenotype of CAR19.20.22 T-cells | Up to 24 months
  Phenotypic analysis of CAR T-cells from blood samples using flow cytometry.
Number of CAR19.20.22 T-cell products manufactured that meet release criteria at Day 8 | At day 8 of manufacturing post-leukapheresis.
  Feasibility will be assessed by counting the number of autologous CAR T-cell products that successfully meet pre-specified release criteria at Day 8 of manufacturing.

CONTACTS AND LOCATIONS:
Overall Officials: Djordje Atanackovic, MD, Principal Investigator — Professor of Medicine
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States